CLINICAL TRIAL: NCT00080834
Title: A Phase II Study Of Oral DJ-927 Administered As A Single Dose Every Three Weeks To Patients With Advanced Or Metastatic Adenocarcinoma Of The Colon Or Rectum
Brief Title: DJ-927 as Second-Line Therapy in Treating Patients With Progressive Locally Advanced or Metastatic Colorectal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000356034; DAIICHI-927A-PRT004; MDA-2003-0749
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; recurrent rectal cancer; stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — tesetaxel

INTERVENTIONS:
Drug: DJ-927

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as DJ-927, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well DJ-927 works as second-line therapy in treating patients with progressive locally advanced or metastatic colorectal adenocarcinoma (cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective tumor response rate in patients with progressive locally advanced or metastatic adenocarcinoma of the colon or rectum treated with DJ-927 as second-line treatment.

Secondary

* Determine the duration of response in patients treated with this drug.
* Determine the time to tumor progression in patients treated with this drug.
* Determine the median survival time in patients treated with this drug.
* Determine the quantitative and qualitative toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to prior first-line treatment regimen (irinotecan-containing vs oxaliplatin-containing).

Patients receive oral DJ-927* on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients receive 1 of 2 selected doses to confirm the previously established maximum tolerated dose

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 56-62 patients (28-31 per stratum) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Progressive locally advanced or metastatic disease
* Received 1 prior irinotecan- or oxaliplatin-containing regimen
* At least 1 measurable lesion

  * Target lesion must be outside field of prior radiotherapy
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* ALT and AST ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Gastrointestinal

* No difficulty with swallowing
* No malabsorption
* No diarrhea (excess of 2-3 stools/day above normal frequency) within the past month
* No history of chronic diarrhea

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No concurrent serious infection
* No other concurrent severe or uncontrolled underlying medical condition that would preclude study participation
* No neuropathy ≥ grade 2
* No history of any severe or life-threatening hypersensitivity reaction
* No psychiatric disorder that would preclude study compliance
* No other malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior myelosuppressive chemotherapy and recovered
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

  * Localized radiotherapy to non-indicator lesions for pain relief allowed provided other methods of pain control are ineffective

Surgery

* At least 4 weeks since prior major surgery and recovered
* No prior major surgery in the stomach or small intestine

Other

* More than 28 days since prior investigational agents (including analgesics and/or antiemetics)
* No other concurrent anticancer therapy
* No other concurrent cytotoxic therapy
* No concurrent grapefruit products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cheverton, MD, ChB, MMED, RadT, Study Chair — Daiichi Pharmaceuticals
Locations (2):
- United States (2):
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - MD Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Result] Rhee JM, Lee FC, Saif MW, et al.: Phase II trial of DJ-927 as a second-line treatment for colorectal cancer demonstrates objective responses. [Abstract] J Clin Oncol 23 (Suppl 16): A-3654, 284s, 2005.